CLINICAL TRIAL: NCT04030104
Title: Imagio® Pivotal Multi-Reader, Multi-Case Study of Optoacoustic Images Versus Imagio® Ultrasound to Guide Decision to Biopsy
Brief Title: Optoacoustic Images Versus Imagio® Ultrasound
Acronym: Reader-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seno Medical Instruments Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: Reader-02 Study
Record Dates: First submitted 2019-05-22; First posted 2019-07-23 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Intervention Model Description: This will be a controlled, blinded, multi-reader, multi-case (MRMC) study using a sequential design. The study will include 15 readers with an additional 5 as back-up readers depending on qualifications and availability. Readers that participated in the Seno PIONEER Study or the Reader-01 Feasibility Study are not eligible to participate as readers in this Pivotal Study.
Who Masked: Outcomes Assessor
Masking Description: Readers will not be provided with information regarding the initial patient diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Imagio IUS (Active Comparator): Read 1 (Control): History + Mammogram (if available) + IUS (Imagio Ultrasound) stills and videos provided), IUS Probability of Malignancy (POM) and Breast Imaging Reporting and Data System (BI-RADS) scored and the data form then locked.
  Interventions: Device: Reader Study - Imagio Ultrasound; Device: Mammography
- Imagio (IUS+OA) (Experimental): Read 2 (Test): History + Mammogram (if available) + IUS (stills and videos provided), and Imagio (IUS+OA) (stills and videos provided). Imagio (IUS+OA) POM and Breast Imaging Reporting and Data System (BI-RADS) assigned after viewing the SenoGram® output. The dataform is locked.
  Interventions: Device: Reader Study Imagio Ultrasound + Optoacoustic Imaging; Device: Mammography

INTERVENTIONS:
Device: Reader Study - Imagio Ultrasound — Imagio ultrasound images to be reviewed as part of Reader study
  Arms: Imagio IUS
Device: Reader Study Imagio Ultrasound + Optoacoustic Imaging — Imagio Ultrasound + Optoacoustic images to be reviewed as part of Reader study
  Arms: Imagio (IUS+OA)
Device: Mammography — Mammography as available per standard of care
  Other Names: Mammo

SUMMARY:
The Imagio® Pivotal Study is intended to evaluate if the results observed in the previous Feasibility Study can be confirmed for pre-specified effectiveness endpoints. Using Intention-to-Diagnose (ITD) masses from the PIONEER Pivotal study, 480 to 840 masses are to be used for the Pivotal Study, the remaining masses will be reserved for training the SenoGram® model.

DETAILED DESCRIPTION:
This will be a controlled, blinded, multi-reader, multi-case (MRMC) study using a sequential design. The study will include 15 readers with an additional 5 as back-up readers depending on qualifications and availability. Readers that participated in the Seno PIONEER Study (NCT01943916) or the Reader-01 Feasibility Study (NCT03708393) are not eligible to participate as readers in this Pivotal Study.

Imagio® [Ultrasound (IUS) + Optoacoustic (OA)] (IUS)(IUS+OA) training will be completed prior to any reads taking place. Read 1 will be immediately followed by Read 2 within the same read session.

ELIGIBILITY:
Inclusion Criteria:

* One analyzable mass per patient: BI-RADS 3 and 4a, 4b, 4c and 5 masses as declared by clinical site investigator via PIONEER study inclusion criteria and categorized as BIRADS 3, 4a, 4b 4c and 5 by conventional diagnostic ultrasound (CDU)
* Masses declared to be in the PIONEER Intention to Diagnose (ITD)/analysis population, including high risk cases per original PIONEER protocol
* Patient age, indication for study entry and available medical history
* Evaluable mammograms and OA and IUS video loops and stills for each mass

Exclusion Criteria:

* Critical missing IUS or OA still image and/or video loop views or incorrect IUS or OA stills and video loops that would preclude a case from being evaluated by readers
* Reader-02 Proficiency Test and training cases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Images from female patients
Enrollment: 480 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-11-03 (Actual); Study Completion 2019-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaan Schaeffer, Study Director — Seno Medical
Locations (1):
- American College of Radiology Center for Research and Innovation, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: New Independent Reader Study (new readers re-reading a sub-set of randomly selected images acquired during PIONEER-01 Study- (NCT01943916)). Reader-02 study execution dates: 30 Jul 2019 to 3 Nov 2019
Pre-assignment Details: Imagio Ultrasound (IUS) and Imagio optoacoustic/ultrasound (IUS+OA) images of breast masses previously acquired from the PIONEER-01 study (NCT01943916) referenced above were used for this study. Reader-02 was a single-arm sequentially read multi reader/case (MRMC) study comparing IUS vs Imagio (IUS+OA). New readers were recruited-NO new subjects/masses. Results were based on biopsy diagnosis or truth panel decision as ground truth obtained during PIONEER-01.
Groups:
- Overall (Subjects Randomly Selected From PIONEER-01 Study): Each subject had one mass that was read by all readers. Each subject served as her own control, with imaging of each mass by both IUS and IUS+OA modalities. Therefore, baseline data are for overall population only.
Period: Overall Study
Arm/Group | Overall (Subjects Randomly Selected From PIONEER-01 Study)
Started | 480
Completed | 480
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-diagnose (ITD)
Groups:
- Overall (Subjects Randomly Selected From PIONEER-01 Study): Each subject had one mass that was read by all readers. Each subject served as her own control, with imaging of each mass by both IUS and IUS+OA modalities. Therefore, baseline data derived from PIONEER-01 for sub set of 480 cases read during Reader-02 Study.
Arm/Group | Overall (Subjects Randomly Selected From PIONEER-01 Study)
Number analyzed (Participants) | 480
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 87
  Not Hispanic or Latino | 387
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 54
  White | 389
  More than one race | 2
  Unknown or Not Reported | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 480
Mass Diagnosis [Count of Participants; unit: Participants] — Mass diagnosis by biopsy result or Truth Panel decision
  Participants
    Subjects (Benign+TPB+HR) | 300
    Subjects (Cancer) | 180

OUTCOME MEASURES:

1. Primary Outcome: Gain in Specificity at Fixed 98% Sensitivity (fSp)
Description: Primary effectiveness endpoint was the difference (gain) in specificity (fSp) at fixed 98% sensitivity for the Imagio IUS+OA relative to IUS alone, across all 15 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth). fSp derived from empirical receiver operating characteristic (ROC) using endpoint interpolation.
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-diagnose (ITD)
Measure: Mean (95% Confidence Interval); unit: % benign+TPB masses correctly identified
Groups:
- IUS Alone: IUS alone imaging
- Imagio (IUS+OA): IUS+OA imaging
Arm/Group | IUS Alone | Imagio (IUS+OA)
Number analyzed (Participants) | 480 | 480
% benign+TPB masses correctly identified | 38.22 [24.85 to 51.59] | 47.20 [35.91 to 58.49]
Statistical Analysis 1: Comparison: IUS Alone vs Imagio (IUS+OA); Test type: Superiority; p = 0.0268, Random Reader, Random Mass — Threshold for statistical significance <0.05; Curve Fitting Method: Empirical

2. Secondary Outcome: Negative Likelihood Ratio (NLR)
Description: NLR for the Imagio IUS+OA relative to IUS alone, across all 15 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth). NLR = [(1-sensitivity) / specificity].
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-diagnose (ITD)
Measure: Mean (95% Confidence Interval); unit: Ratio
Groups:
- Imagio Alone: IUS alone imaging
Arm/Group | Imagio Alone | Imagio (IUS+OA)
Number analyzed (Participants) | 480 | 480
Ratio | 0.053 [0.037 to 0.070] | 0.047 [0.032 to 0.062]

3. Secondary Outcome: Positive Likelihood Ratio (PLR)
Description: PLR for the Imagio IUS+OA relative to IUS alone, across all 15 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth). PLR = [sensitivity / (1-specificity)].
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Total population of subjects/masses
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | IUS Alone | Imagio (IUS+OA)
Number analyzed (Participants) | 480 | 480
Ratio | 1.548 [1.498 to 1.597] | 1.959 [1.870 to 2.051]

4. Secondary Outcome: Partial Area Under the Curve (pAUC)
Description: pAUC considers only the region of the area under the ROC curve that corresponds to clinically relevant values of sensitivity, defined as 95% to 100%, for Imagio IUS+OA vs. IUS alone, averaged across 15 readers. Both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth). A higher pAUC indicates better diagnostic accuracy.
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-diagnose (ITD)
Measure: Mean (95% Confidence Interval); unit: Percentage of Probability
Arm/Group | IUS Alone | Imagio (IUS+OA)
Number analyzed (Participants) | 480 | 480
Percentage of Probability | 0.0205 [0.0191 to 0.0219] | 0.0244 [0.0230 to 0.0258]

ADVERSE EVENTS:
Time Frame: Baseline to 12 months +/- 30 days follow-up
Groups:
- Overall (Subjects Randomly Selected From PIONEER-01 Study): Each subject had one mass that was read by all readers. Each subject served as her own control, with imaging of each mass by both IUS and IUS+OA modalities. Therefore, safety data are for overall population only.
Arm/Group | Overall (Subjects Randomly Selected From PIONEER-01 Study)
All-Cause Mortality (participants affected / at risk) | 0/480
Serious Adverse Events (participants affected / at risk) | 2/480
Other Adverse Events (participants affected / at risk) | 14/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (Subjects Randomly Selected From PIONEER-01 Study) (N=480)
Device breakage (General disorders) | 1 (1) — Right saline breast implant rupture
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Non-small cell lung cancer Stage I
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (Subjects Randomly Selected From PIONEER-01 Study) (N=480)
Paraesthesia (Nervous system disorders) | 5 (5) — Tingling sensation
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Post-procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study are the property of Seno Medical Instruments, Inc. All publications (manuscripts, abstracts or other modes of presentation) must be submitted and reviewed and approved in writing by Seno Medical Instruments, Inc., in advance of submission. The over all study results will first be submitted as a primary paper.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT04030104/Prot_SAP_001.pdf